CLINICAL TRIAL: NCT03721757
Title: NICO - CA209-891: Neoadjuvant and Adjuvant Nivolumab as Immune Checkpoint Inhibition in Oral Cavity Cancer
Brief Title: CA209-891: Neoadjuvant and Adjuvant Nivolumab as Immune Checkpoint Inhibition in Oral Cavity Cancer
Acronym: NICO
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The Clatterbridge Cancer Centre NHS Foundation Trust (Other)
Collaborators: University of Liverpool (Other); Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: C0947; 2017-005015-13 (EudraCT Number); ISRCTN17428671 (Registry Identifier: ISRCTN); CA209-891 (Other Grant/Funding Number: Bristol Myers Squibb)
Record Dates: First submitted 2018-07-23; First posted 2018-10-26 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Squamous Cell Carcinoma of the Oral Cavity
Keywords: Head and Neck cancer; Squamous cell carcinoma
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Head and Neck Neoplasms; Carcinoma, Squamous Cell | interventions — Nivolumab; Surgical Procedures, Operative; Radiotherapy; Radiotherapy, Adjuvant; Chemoradiotherapy; Chemoradiotherapy, Adjuvant

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nivolumab, Surgery, Radiotherapy (Other): Patients will be treated with a single dose of nivolumab (240mg flat dose), followed by surgery to remove their tumour within 1-2 weeks.
  Based on pathological risk factors determined following surgery, patients will be assigned to undergo adjuvant radiotherapy or chemoradiotherapy. Patients with low risk criteria following surgery will be assigned to radiotherapy.
  A single dose of nivolumab (240mg flat dose) will be given between surgery and commencement of radiotherapy (1-2 weeks prior).
  Radiotherapy will be administered over 30 fractions i.e. over 30 days (Monday to Friday for 6 consecutive weeks).
  Following completion of radiation (within 1-2 weeks), patients will commence adjuvant nivolumab, with a total of 6 doses (480mg flat dose) given at 4 weekly intervals
  Interventions: Biological: Nivolumab, Surgery, Radiotherapy
- Nivolumab, Surgery, Chemoradiotherapy (Other): Patients will be treated with a single dose of nivolumab (240mg flat dose), followed by surgery to remove their tumour within 1-2 weeks.
  Based on pathological risk factors determined following surgery, patients will be assigned to undergo adjuvant radiotherapy or chemoradiotherapy. Patients with high risk criteria following surgery will be assigned to chemoradiotherapy.
  A single dose of nivolumab (240mg flat dose) will be given between surgery and chemoradiotherapy (1-2 weeks prior).
  Chemoradiotherapy will be administered over 30 fractions i.e. over 30 days with concomitant Cisplatin (100mg/m2) on day 1 and 21.
  Following completion of radiation (within 1-2 weeks), patients will commence adjuvant nivolumab, with a total of 6 doses (480mg flat dose) given at 4 weekly intervals.
  Interventions: Biological: Nivolumab, Surgery, Chemoradiotherapy

INTERVENTIONS:
Biological: Nivolumab, Surgery, Radiotherapy — A single dose of nivolumab 7-14 days before curative surgery. A further single dose will be administered following surgery and prior to radiotherapy commencing. Six further doses of nivolumab will be received post radiotherapy
  Other Names: Curative Surgery; Adjuvant Radiotherapy
  Arms: Nivolumab, Surgery, Radiotherapy
Biological: Nivolumab, Surgery, Chemoradiotherapy — A single dose of nivolumab 7-14 days before curative surgery. A further single dose will be administered following surgery and prior to Chemoradiotherapy (cisplatin) commencing. Six further doses of nivolumab will be received post radiotherapy
  Other Names: Curative surgery; Adjuvant chemoradiotherapy
  Arms: Nivolumab, Surgery, Chemoradiotherapy

SUMMARY:
This trial is to investigate the use of nivolumab in sequence with standard of care surgery and radiation/chemoradiation in locally advanced oral cavity Squamous cell carcinoma of the oral cavity.

DETAILED DESCRIPTION:
Squamous cell carcinoma of the oral cavity is usually treated with surgery, often followed by radiation therapy with or without chemotherapy. Unfortunately despite this treatment, it recurs or spreads in about half of patients. In this trial the investigators aim to investigate the use of nivolumab in sequence with standard of care surgery and radiation/chemoradiation.

Following confirmation of eligibility patients will be treated with a single dose of nivolumab 1-2 weeks prior to surgery to remove their tumour. Based on pathological risk factors determined following surgery, patients will be assigned to undergo adjuvant radiotherapy or chemoradiotherapy. Patients with high risk criteria (Extra capsular spread, involved margins) will be assigned to chemoradiotherapy. A further single dose of nivolumab will be given between surgery and commencement of radiotherapy or chemoradiotherapy.

Following completion of chemo/radiation, patients will commence adjuvant nivolumab, with a total of 6 doses given at 4 weekly intervals. Patients will be followed up for 12 months post surgery.

The primary objectives of this trial is to determine disease free survival at 12 months post surgery and the feasibility of recruiting to both cohorts.

ELIGIBILITY:
1. Signed, written informed consent
2. Subjects must be willing and able to comply with scheduled visits and procedures
3. Histologically confirmed squamous cell carcinoma of the oral cavity, (oral tongue (anterior 2/3), gingiva/alveolus, floor of mouth, buccal sulcus, retromolar trigone, and hard palate as defined by ICD-10 codes)
4. Subjects willing to have a fresh biopsy performed, or archival tissue available from diagnostic biopsy meeting requirements set out in laboratory manual.
5. Clinically and/or radiologically staged as T1-4 N1-3 or any T3-4 N0 (unless T4 on the basis of bone invasion only). Staging based upon the AJCC/UICC TNM 8th Edition.
6. Surgery planned as primary treatment modality with patients fit for major resection ± reconstruction surgical procedure.
7. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
8. 18 years or over at time of provision of consent for trial inclusion.
9. Screening laboratory values must meet the following criteria

   * WBC ≥ 2000/µL
   * Neutrophils ≥ 1500/uL
   * Platelets ≥ 100x103/uL
   * Hemoglobin ≥ 9.0 g/dL
   * Serum creatinine ≤ 1.5 x ULN or calculated creatinine clearance > 40 mL/min (using the Cockcroft-Gault formula)
   * AST ≤ 3.0 x ULN
   * ALT ≤ 3.0 x ULN
   * Total Bilirubin ≤ 1.5 x ULN (except subjects with Gilbert Syndrome who must have a total bilirubin level of < 3.0x ULN).
10. Women of childbearing potential (WOCBP) must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) within 24 hours prior to the start of study drug.
11. Women must not be breastfeeding
12. WOCBP must agree to follow instructions for method(s) of contraception for a period of 30 days (duration of ovulatory cycle) plus the time required for the investigational drug to undergo approximately five half-lives. WOCBP randomized/assigned to receive nivolumab should use an adequate method to avoid pregnancy for 5 months (30 days plus the time required for nivolumab to undergo approximately five half-lives) after the last dose of investigational drug.
13. Males who are sexually active with WOCBP must agree to follow instructions for method(s) of contraception for a period of 90 days (duration of sperm turnover) plus the time required for the investigational drug to undergo approximately five half-lives
14. Males randomized to receive nivolumab who are sexually active with WOCBP must continue contraception for 7 months (90 days plus the time required for nivolumab to undergo approximately five half-lives) after the last dose of investigational drug. Azoospermic males and WOCBP who are continuously not heterosexually active are exempt from contraceptive requirements. However they must still undergo pregnancy testing as described in these sections. Investigators shall counsel WOCBP and male subjects who are sexually active with WOCBP on the importance of pregnancy prevention and the implications of an unexpected pregnancy Investigators shall advise WOCBP and male subjects who are sexually active with WOCBP on the use of highly effective methods of contraception. Highly effective methods of contraception which have a failure rate of < 1% when used consistently and correctly

Exclusion Criteria:

1. Tumours staged as T4 on the basis of bone invasion only and in the absence of nodal metastases.
2. Distant metastases detected, or suspected on imaging
3. Unfit for chemoradiotherapy, due to comorbidity.
4. Previous malignancy requiring treatment within the last 3 years (with the exception of non-melanoma skin cancers, and the following in situ cancers: bladder, gastric, colon, oesophageal endometrial, cervical/dysplasia, melanoma, or breast). Prior head and neck cancer within the last three years is allowed if the tumour was treated with surgery only, and did not require radiotherapy.
5. Prior head and neck radiotherapy
6. On immunosuppressive medication (including steroids at dose equivalent to prednisolone >10mg/day unless used as replacement therapy).
7. Subjects with an active, known or suspected autoimmune disease. Subjects with type I diabetes mellitus, hypothyroidism only requiring hormone replacement, skin disorders (such as vitiligo, psoriasis, or alopecia) not requiring systemic treatment, lichen planus or other conditions not expected to recur in the absence of an external trigger are permitted to enrol.
8. Known human immunodeficiency virus (HIV) or viral hepatitis infection.
9. Women who are pregnant or breastfeeding
10. Known medical condition that, in the investigator's opinion, would increase the risk associated with study participation or study drug administration or interfere with the interpretation of safety results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2019-05-10 (Actual); Primary Completion 2025-02-24 (Actual); Study Completion 2025-02-24 (Actual)

PRIMARY OUTCOMES:
Disease free survival | Patients will be followed up for 12 months following surgery
  1 year disease free survival defined as disease recurrence or death at 12 months from surgery
Recruitment Rate | Period of recruitment
  Measured as the number of patients/site/month

SECONDARY OUTCOMES:
Overall survival | Patients will be followed up for 12 months following surgery
  Overall survival measured as the time from surgery to death by any cause
Surgical complications - Infection rate | up to 8 weeks post date of surgery
  Measured as incidence of post surgical infection
Surgical complications - length of hospital admission | up to 8 weeks post date of surgery
  Measured as length of time between admission for surgery and discharge
Surgical complications - free flap failure | up to 8 weeks post date of surgery
  Measured as incidence of failure of free flap reconstruction
Surgical complications - perioperative (30-day mortality) | up to 30 days post date of surgery
  Measured as Incidence of death post surgery by any cause
Assessment of adverse events | Following participants informed consent up to 100 days following last dose of trial treatment.
  Assessment of adverse events, adverse events recorded will be classified using CTCAE v4
The change of Quality of Life: EORTC QLQ-C30 v3 | Patients will be followed up for 12 months following surgery
  The change of quality of life is measured using the EORTC QLQ-C30 v3 quality of life questionnaire. The quality of life scale is transformed into a score of 0 to 100, derived by a 4-point Likert scale. A higher score represents a higher level of quality of life.
The change of symptom | Patients will be followed up for 12 months following surgery
  The change of symptoms is measured using the EORTC quality of life questionnaire (EORTC QLQ) Head and Neck cancer module (QLQ-H&N35). The symptom scale is transformed into a score of 0 to 100, derived by a 4-point Likert scale. A higher score represents a higher level of symptom.

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Sacco, MBChB, Principal Investigator — University of Liverpool
Locations (1):
- Clatterbridge Cancer Centre NHS Foundation Trust, Bebington, United Kingdom

IPD SHARING:
Plan to Share IPD: No